CLINICAL TRIAL: NCT03840837
Title: Cholinergic Neurotransmission - A Common Underlying Mechanism of Cognitive and Gait Impairment in Parkinson Disease
Brief Title: Cholinergic Neurotransmission in Mobility and Cognition in Parkinson Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, F. Rainer von Coelln, MD, Assistant Professor, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HP-00084074; 3P30AG028747-13S3 (NIH)
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Parkinson Disease; Parkinson Disease Dementia
Keywords: cognitive impairment; Parkinson disease dementia; wearable sensor; gait analysis; rivastigmine; cholinesterase inhibitor
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: All participants perform a baseline assessment (arm 1 - cross-sectional). A subgroup of participants (based on physician and participant choice) proceed to a 12-week treatment phase with the study drug (transdermal rivastigmine) and subsequent follow-up assessment (arm 2 - longitudinal).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm 1: baseline only (cross-sectional) (No Intervention): At baseline, all participants will undergo instrumented gait/balance testing, using a wearable sensor (Dynaport MT), and cognitive testing, using a computerized cognitive test battery (NeuroTrax Mild Cognitive Impairment & Early Dementia Battery by MindStreams). In other words, all participants will be part of arm 1.
- Arm 2: rivastigmine (longitudinal) (Experimental): As study intervention, a subgroup of participants will then be treated with transdermal rivastigmine patch for 12 weeks, with dose increases every 4 weeks and titration up to 13.3 mg/24h, if tolerated. For the arm 2 subgroup of participants, the same assessment that was performed at baseline (quantitative gait testing and NeuroTrax computerized cognitive test battery) will be repeated after 12 weeks, with the patient on a stable dose of transdermal rivastigmine.
  Interventions: Drug: Rivastigmine transdermal patch

INTERVENTIONS:
Drug: Rivastigmine transdermal patch — Titration of transdermal rivastigmine, as per arm description.
  Other Names: Exelon transdermal patch
  Arms: Arm 2: rivastigmine (longitudinal)

SUMMARY:
This is a single-site non-randomized open label pilot study. The investigators will use accelerometer-based instrumented gait analysis and computerized cognitive testing to study the interaction of motor and cognitive dysfunction in Parkinson disease dementia (PDD), and the effect of rivastigmine on motor and cognitive performance. All study participants will be tested for motor and cognitive performance at baseline (arm 1). A subgroup of study participants will then be treated with rivastigmine for 12 weeks (arm 2), and the effect of this treatment on gait measures and cognitive measures will be analyzed at the follow-up visit 12 weeks after the baseline visit. Specifically, we will determine which components of motor and cognitive impairment are associated with each other, and which components of the two domains respond to rivastigmine-mediated stimulation of cholinergic neurotransmission.

DETAILED DESCRIPTION:
This is a single-site non-randomized open label clinical trial in patients with Parkinson disease (PD) and mild to moderate cognitive deficits, designed to 1) identify associations between cognitive impairment and gait impairment, and 2) identify cognitive domains and gait measures that improve after 12 weeks of treatment with rivastigmine. Aim 1 will be addressed with a cross-sectional approach (arm 1, baseline only, all participants), and aim 2 will be addressed with a longitudinal interventional approach (arm 2, 12 week-treatment with rivastigmine, subgroup of participants).

Patients with idiopathic Parkinson disease (PD) and mild to moderate cognitive deficits amounting to PD dementia (PDD) will be enrolled. At baseline (arm 1), all participants will perform the timed-up-and-go test (TUG), wearing a light-weight sensor device strapped to the lower back with a neoprene belt. Participants will also complete a computerized cognitive test battery (NeuroTrax Mild Cognitive Impairment & Early Dementia Battery by MindStreams). A subgroup of participants (arm 2) will then be treated with transdermal rivastigmine for 12 weeks, with dose increases every 4 weeks and titration up to 13.3 mg/24h, if tolerated. The same assessment (quantitative gait testing and NeuroTrax computerized cognitive test battery) will be repeated after 12 weeks, with the participant on a stable dose of transdermal rivastigmine.

The investigators will analyze correlation of iTUG measures and cognitive measures at baseline (cross-sectional analysis). The investigators will also analyze change in iTUG measures and cognitive measures between baseline and follow-up for the subgroup of participants in arm 2 (in other words, before and after rivastigmine treatment; longitudinal analysis).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Diagnosis of idiopathic Parkinson disease.
* Mild to moderate cognitive impairment, as determined by a MoCA score of ≤ 25 and ≥ 10.
* Patient passes the Evaluation to Sign Consent (ESC) or a legally authorized representative (LAR) is present at the time of enrollment and signs the informed consent form on behalf of the patient.
* Patient is enrolled (or willing to be enrolled) in the University of Maryland Parkinson Disease and Movement Disorders Center PD Research Database (HP 42195)

Exclusion Criteria:

* Advanced Parkinson disease (Hoehn & Yahr stage 5), with inability to walk unassisted.
* Other medical condition(s) that significantly interfere(s) with gait and balance (e.g., advanced arthritis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Timed-Up-and-Go (TUG) duration [s] | Data analysis will be completed within 6 months of completing study enrollment.
  Time participant needs to complete the TUG.
NeuroTrax Executive Function score | Data analysis will be completed within 6 months of completing study enrollment.
  Result of the NeuroTrax computerized cognitive test of executive function.

CONTACTS AND LOCATIONS:
Overall Officials: Rainer von Coelln, Dr. med., Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland School of Medicine, Dept. of Neurology, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
All data generated during this project will be shared with the scientific community through peer-reviewed publications and presentations at national and international conferences.
  We will share our raw data with qualified collaborating scientists upon request. Only aggregated data of study participants will be made available to other researchers.